CLINICAL TRIAL: NCT05667987
Title: Evaluation of the Benefit of Lidocaine on the Prevention of the Risk of Post Endoscopic Retrograde Cholangio-pancreatography Pancreatitis.
Acronym: PEPLID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-A01658-35
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: ERCP Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia without intravenous lidocaine administration (No Intervention)
- General anesthesia with intravenous lidocaine administration (Experimental)
  Interventions: Drug: Intravenous lidocaine administration

INTERVENTIONS:
Drug: Intravenous lidocaine administration — General anesthesia with intravenous lidocaine administration
  Arms: General anesthesia with intravenous lidocaine administration

SUMMARY:
The goal of this study is, in a population of patients undergoing ERCP surgery, treated preventively with NSAIDs and divided into two groups according to the absence (group 1) or presence (group 2) of intravenous lidocaine in the general anesthesia protocol.

The main objective of this study is to compare the incidence of post-ERCP pancreatitis between the two groups.

type of study: clinical trial participant population/health conditions: Patients with ERCP surgery

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized, single-blind study of two parallel groups of patients undergoing ERCP surgery

* Group 1 (n=900): General anesthesia without IV lidocaine administration
* Group 2 (n=900): General anesthesia with IV lidocaine administration

Randomization Patients who have given written informed consent and received confirmation of eligibility will be randomized into the study according to a randomization list. According to the randomization, patients will be divided into two equal groups of 900 patients (anesthesia with and without lidocaine). The randomization list will be established by a centralized computer procedure.

PAP prevention protocols Treatment with indomethacin (100mg intrarectally), which is the reference preventive treatment, will be administered systematically in both groups just before anesthesia (or during anesthesia if ERCP is preceded by an echo-endoscopy). The endoscopic techniques to prevent PAP (pancreatic prosthesis, double guide wire technique, infundibulotomy, needle pre-cutting ...) will be used by the operator according to his procedural habits and will be reported in the CRF.

Anesthesia protocol

All patients will be operated under general anesthesia with orotracheal intubation without premedication with the same anesthesia protocol:

At induction: a hypnotic (propofol or hypnomidate) combined with a morphine (sufentanil or remifentanyl) and low doses of Ketamine and midazolam, with or without curarization.

In maintenance phase sevoflurane. Blood pressure will be maintained by administration of ephedrine, neosynephrine or baby noradrenaline. The patient's hydration will be ensured by an infusion of Ringer Lactate (20ml/Kg).

In the postoperative period, analgesic treatment will be systematically administered with, according to the needs, palliative analgesics 1 or 2 or morphine titration.

Lidocaine administration protocol Patients randomized in group 2 will receive during anesthesia a treatment with 1% non-adrenalized Lidocaine.

An initial bolus (1.5mg/kg) will be administered at induction of anesthesia (or upon ERCP decision if echo-endoscopy is in progress).

Then IVSE of lidocaine at 2mg/Kg/hr will be started for one hour (to be continued in the ICU if needed).

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient who has read and signed the consent form for participation in the study
* Patient candidate for ERCP with virgin papilla

Exclusion Criteria:

* Patient with sphincterotomized papilla
* Patient under court protection, guardianship or curatorship
* Pregnant woman or woman of childbearing age without highly effective contraception for the duration of the study (surgically sterile, intrauterine device (> 14 days), hormonal contraception (same dose and formulation for at least 6 months), sexual abstinence. Women after menarche and until they become postmenopausal, unless they are permanently infertile or have undergone surgical sterilization, are considered to be of childbearing age, i.e. fertile. A postmenopausal condition is defined as the absence of menstruation for 12 months without any other medical cause
* Patient not affiliated with the French social security system
* Patient participating in another clinical research protocol
* Impossibility to give the subject informed information and/or written informed consent: dementia, psychosis, disorders of consciousness, non-French speaking patient
* Contraindication to the use of NSAIDs
* Contraindication to anesthesia or to the administration of any of the products used in anesthesia protocols (including lidocaine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-01-18 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Plasma lipase level | Hour 24
  A plasma lipase level greater than or equal to 3N, considered to be indicative of a PAP, is the primary endpoint of the study

SECONDARY OUTCOMES:
Abdominal pain intensity | Hour 24
  Assessment of abdominal pain on a simple numerical scale
Pancreatic ultrasound or CT scan data | Hour 24
  Pancreatic ultrasound or CT scan data if available
Severity of pancreatitis | Hour 24
  Severity of pancreatitis according to the ATLANTA 2012 criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé des Peupliers, Paris, France

IPD SHARING:
Plan to Share IPD: No